CLINICAL TRIAL: NCT00856193
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center, Two-period Crossover Study to Investigate the Bronchodilatory Effect of 50 µg NVA237 Inhaled Once Daily in Patient With Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: A Study to Investigate the Bronchodilatory Effect of NVA237 in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CNVA237A2207; 2008-006849-28 (EudraCT Number)
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Bronchodilator
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo then NVA237 50μg (Placebo Comparator): Placebo 50 μg capsules followed by NVA237 50 μg capsules for inhalation once daily with Concept 1 device.
  Interventions: Drug: Placebo; Drug: NVA237
- NVA237 50μg then placebo (Experimental): NVA237 50 μg capsules followed by matching placebo 50 μg capsules for inhalation once daily with Concept 1 device.
  Interventions: Drug: Placebo; Drug: NVA237

INTERVENTIONS:
Drug: Placebo — Matching placebo capsules were supplied for inhalation once daily with Concept 1 device.
Drug: NVA237 — NVA237 50 μg capsules were supplied for inhalation once daily with Concept 1 device.

SUMMARY:
This study was intended to assess how well inhaled NVA237 opens up the airways of patients with mild, moderate or severe COPD over a 24 hour period after a 14 day treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged greater than 40 years with COPD Current or ex-smokers

Exclusion Criteria:

* Cardiac (heart) disorders, history of asthma, requiring oxygen therapy. Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Spartanburg Medical Research, Spartanburg, South Carolina, United States
- Harrison Clinical Research Deutschland GmbH, Albrechtstrasse 14, Munich, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were randomized into one of two sequences to receive either NVA237 50 μg followed by placebo or placebo followed by NVA237 50 μg.
Groups:
- Placebo Then NVA237 50μg: Placebo 50 µg capsules followed by NVA237 50 µg capsules for inhalation once daily with Concept 1 device.
Period: Period 1
Arm/Group | NVA237 50μg Then Placebo | Placebo Then NVA237 50μg
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0
Period: Period 2
Arm/Group | NVA237 50μg Then Placebo | Placebo Then NVA237 50μg
Started | 16 | 17
Completed | 16 | 15
Not Completed | 0 | 2
Not completed — Abnormal test procedure results | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Patients: NVA237 50 μg capsules for inhalation once daily with Concept 1 device. Matching placebo 50 µg capsules for inhalation once daily with Concept 1 device.
Arm/Group | All Randomized Patients
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (9.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve (AUC) 0-24 Hours on Day 14
Description: Forced Expiratory Volume in one second (FEV1) was calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. This outcome measures the change is FEV1 from predose (day 1) to the readings taken 0-24 hours post dose on day 14. The variable was analyzed with an analysis-of-covariance model which included baseline FEV1 value as a covariate.
Time Frame: From Day 1 to 0-24 hours after drug administration on Day 14
Population: Efficacy analysis set
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- NVA237 50μg: NVA237 50 μg capsules were supplied by Novartis for inhalation once daily with Concept 1 device.
- Placebo: Matching placebo capsules were supplied by Novartis for inhalation once daily with Concept 1 device.
Arm/Group | NVA237 50μg | Placebo
Number analyzed (Participants) | 31 | 32
Liters | 1.827 (0.0330) | 1.664 (0.0324)

2. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) AUC 0-12 Hours on Day 14
Description: Forced Expiratory Volume in one second (FEV1) was calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. This outcome measures the change is FEV1 from pre-dose (day 1) to the readings taken 0-12 hours post dose on day 14. The variable was analyzed with an analysis-of-covariance model which included baseline FEV1 value as a covariate.
Time Frame: From day 1 to 0 -12 hours after drug administration on Day 14
Population: Efficacy analysis set
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 50μg | Placebo
Number analyzed (Participants) | 31 | 32
Liters | 1.879 (0.0346) | 1.714 (0.0340)

3. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) AUC 12-24 Hours on Day 14
Description: Forced Expiratory Volume in one second (FEV1) was calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. This outcome measures the change is FEV1 from pre-dose (day 1) to the readings taken 12-24 hours post dose on day 14. The variable was analyzed with an analysis-of-covariance model which included baseline FEV1 value as a covariate.
Time Frame: From Day 1 to 12 hours-24 hours after drug administration on Day 14
Population: Efficacy analysis set
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 50μg | Placebo
Number analyzed (Participants) | 31 | 32
Liters | 1.776 (0.0344) | 1.615 (0.0339)

4. Secondary Outcome: Number of Participants Who Experienced Adverse Events (AEs), Serious Adverse Events (SAEs)
Description: According to FDA 21CFR 314.80, a serious adverse event (SAE) is described as any adverse event that leads to death, is life threatening , causes or prolongs hospitalization, results in a congenital anomaly, or any other important medical event not described above. See Adverse Events module for details.
Time Frame: Day 14
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | NVA237 50μg | Placebo
Number analyzed (Participants) | 31 | 33
Participants
  Overall Adverse Events | 2 | 4
  Serious Adverse Events (SAEs) | 0 | 0

ADVERSE EVENTS:
Groups:
- NVA237 50 μg: NVA237 50 μg capsules were supplied by Novartis for inhalation once daily with Concept 1 device.
Arm/Group | Placebo | NVA237 50 μg
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/31
Other Adverse Events (participants affected / at risk) | 2/33 | 0/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=33) | NVA237 50 μg (N=31)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.